CLINICAL TRIAL: NCT00306254
Title: A Phase 2B, Randomized, Multicenter, Dose-Ranging Study Assessing the Safety and Efficacy of PD 0348292 in the Prevention of Venous Thromboembolic Events (VTE) in Subjects Undergoing an Elective, Unilateral Total Knee Replacement
Brief Title: Evaluation of PD 0348292 for Preventing Blood Clots in the Lungs or Deep Leg Veins of Patients After Knee Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A5571010
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — N-(4-chlorophenyl)-N-(2-fluoro-4-(2-oxopyridin-1(2H)-yl)phenyl)-4-methoxypyrrolidiine-1,2-dicarboxamide; Enoxaparin

INTERVENTIONS:
Drug: PD 0348292
Drug: Enoxaparin

SUMMARY:
To study the safety and effectiveness of several doses of PD 0348292 compared to enoxaparin in preventing blood clots in the lungs or deep leg veins of patients after knee surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women scheduled for an elective, unilateral total knee replacement who are otherwise healthy.

Exclusion Criteria:

* History of deep vein thrombosis or pulmonary embolism, suspected postthrombotic state, bleeding or clotting disorders, or cardiovascular, renal or liver disease within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225
Dates: Start 2006-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the incidence of total venous thromboembolism (including all proximal and distal deep vein thrombosis [DVT] and pulmonary embolism [PE])
The primary safety endpoint is the incidence of total bleeding.

SECONDARY OUTCOMES:
Secondary efficacy endpoints are incidence of proximal DVT, distal DVT, and PE.
Secondary safety endpoints are incidence of major and minor bleeding, all-cause mortality, abnormal liver function test elevation, adverse events and serious adverse events, and changes in clinical laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (100):
- United States (32):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, North Little Rock, Arkansas
  - Pfizer Investigational Site, Encinitas, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
- Australia (11):
  - Pfizer Investigational Site, Caringbah, New South Wales
  - Pfizer Investigational Site, Kogarah, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Daw Park, South Australia
  - Pfizer Investigational Site, Box Hill, Victoria
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Dandenong, Victoria
  - Pfizer Investigational Site, East Bentleigh, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
  - Pfizer Investigational Site, West Perth, Western Australia
- Canada (10):
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Guelph, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Thunder Bay, Ontario
  - Pfizer Investigational Site, Weston, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Santiago, RM, Chile
- Colombia (4):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Floridablanca, Santander Department
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Czechia (9):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Chomutov
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Jihlava
  - Pfizer Investigational Site, Kladno
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Třebíč
  - Pfizer Investigational Site, Uherské Hradiště
- Denmark (7):
  - Pfizer Investigational Site, Hellerup
  - Pfizer Investigational Site, Hoersholm
  - Pfizer Investigational Site, Hvidovre
  - Pfizer Investigational Site, Kjellerup
  - Pfizer Investigational Site, Kolding
  - Pfizer Investigational Site, Silkeborg
  - Pfizer Investigational Site, Viborg
- France (2):
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
- Italy (3):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Piacenza
- Poland (6):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bytom
  - Pfizer Investigational Site, Piekary Śląskie
  - Pfizer Investigational Site, Sosnowiec
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Parede
  - Pfizer Investigational Site, Setúbal
- Russia (3):
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Samara
  - Pfizer Investigational Site, Yaroslavl
- Pfizer Investigational Site, Košice, Slovakia
- South Africa (2):
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
- Spain (4):
  - Pfizer Investigational Site, Barcelona, BARCELONA
  - Pfizer Investigational Site, Alcorcón, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Mirasierra, Madrid
- United Kingdom (2):
  - Pfizer Investigational Site, Epsom, Surrey
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5571010&StudyName=Evaluation%20of%20PD%200348292%20for%20preventing%20blood%20clots%20in%20the%20lungs%20or%20deep%20leg%20veins%20of%20patients%20after%20knee%20surgery